CLINICAL TRIAL: NCT06190730
Title: REmote Symptom COllection to improVE postopeRative Care
Acronym: RECOVER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00007172
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-01

CONDITIONS: Gastrointestinal Cancer; Gastrointestinal Tumor; Gastrointestinal Tumor Surgery; Gastrointestinal Surgery
Keywords: speech system; large language model; ai
MeSH Terms: conditions — Gastrointestinal Neoplasms; Digestive System Neoplasms

STUDY DESIGN:
Intervention Model Description: The Voice-Assisted Remote Symptom Monitoring System (VARSMS) will be installed on Amazon Echo Dot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Besides the consent process, subjects in this arm will have no other research-specific activities until after 40 days after the surgery for an exit interview.
- Voice-Assisted Remote Symptom Monitoring System (VARSMS) group (Experimental): Subjects in this group will be issued the device, to be activated 1 day after discharge. The device will administer a set of questions daily.
  Interventions: Other: Voice-Assisted Remote Symptom Monitoring System (VARSMS)

INTERVENTIONS:
Other: Voice-Assisted Remote Symptom Monitoring System (VARSMS) — Utilizing an Alexa Skill activated via an Amazon Echo Dot device, this system will administer two patient-reported outcomes measures to subjects. This will not be used as basis for diagnosis, nor for any clinical intervention.
  Other Names: Voice-Assisted Remote Symptom Monitoring System (VARSMS)- customization phase
  Arms: Voice-Assisted Remote Symptom Monitoring System (VARSMS) group

SUMMARY:
There are vulnerabilities in post-discharge care transition for patients after undergoing resection of malignant gastrointestinal tumors. This study aims to investigate the possibility of utilizing Voice-Assisted Remote Symptom Monitoring System (VARSMS) to alleviate some of these challenges.

DETAILED DESCRIPTION:
Randomized controlled trial comparing post-op patients randomized to using the VARSMS vs control.

ELIGIBILITY:
Inclusion criteria

1. At least 18 years old. Ages of subjects >89 will simply be reported as >90.
2. Scheduled for a GI surgery for management of a tumor in a participating hospital.
3. Fluent in oral and written English.
4. Has consistent and continued full access to an operational Wi-Fi for the duration of the study.

Exclusion criteria

1. Unable to provide informed consent.
2. Not willing to commit to regular participation in the study to include daily use (40 days) of the study application.
3. Life expectancy of less than 60 days.
4. In the opinion of the investigator, participation in this study is contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Custom questionnaire based on NCI PRO CTCAE (National Cancer Institute- Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events) | 40 days
  Daily symptom-based self-reported assessment on dyspnea, fever, melena, pain, wound healing, activities of daily living, sensorium, gastrointestinal motility, dysphagia, pitting edema, mood, and an option to mention symptoms not asked of.
  This is monitored by the research team, and any concerning finding, at the discretion of the site's physician, will be relayed to the subject's treating physician.
  Treating physician has final decision on whether to address referral by adjustment of management.

SECONDARY OUTCOMES:
SASSI (Subjective Assessment of Speech System Interfaces) | 40 days
  After interacting with the speech system for 40 days from the day after discharge, this questionnaire assesses the patient on their experience, having them rate the system based on system response accuracy, likeability, cognitive demand, annoyance, habitability, and speed.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - MedStar Health, Baltimore, Maryland
  - Creighton University, Omaha, Nebraska